CLINICAL TRIAL: NCT00099697
Title: Biologic Effects of DHEA in Humans
Brief Title: Biologic Effects of Dehydroepiandrosterone (DHEA) in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: AG0013; 5P60AG013629 (NIH); 5R01AG020076 (NIH); 5K23RR016191 (NIH); 3P30DK056341 (NIH); 5P60DK020579 (NIH); 2M01RR000036 (NIH)
Record Dates: First submitted 2004-12-17; First posted 2004-12-20 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2004-12

CONDITIONS: Aging; Obesity; Insulin Resistance
Keywords: abdominal fat; dehydroepiandrosterone; Insulin sensitivity
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Dehydroepiandrosterone

INTERVENTIONS:
Drug: DHEA

SUMMARY:
The purpose of this study is to determine whether DHEA replacement therapy decreases abdominal fat and improves insulin sensitivity.

DETAILED DESCRIPTION:
Studies on rats and mice have shown that the adrenal hormone dehydroepiandrosterone (DHEA) reduces abdominal visceral fat and protects against insulin resistance. This study was done to learn if DHEA replacement therapy decreases abdominal obesity and improves insulin action in humans.

Participants were randomly assigned to receive 50 mg per day of DHEA or a placebo at bedtime for 6 months. Participants underwent magnetic resonance imaging (MRI) and oral glucose tolerance tests at the beginning and conclusion of the study. Other tests included measurements of hormones and lipids.

ELIGIBILITY:
Inclusion Criteria:

* 65 to 78 years old
* Physically healthy
* Non-smoker
* On stable medications for at least 6 months
* Stable body weight for the past year

Exclusion Criteria:

* Serious active medical problems
* Hormone therapy
* Abnormal PSA (prostate specific antigen) in men

Ages: 65 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 56
Dates: Start 2001-06; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
6-month change in visceral and subcutaneous abdominal fat

CONTACTS AND LOCATIONS:
Overall Officials: John O. Holloszy, MD, Principal Investigator — Washington University School of Medicine; Dennis T. Villareal, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Hansen PA, Han DH, Nolte LA, Chen M, Holloszy JO. DHEA protects against visceral obesity and muscle insulin resistance in rats fed a high-fat diet. Am J Physiol. 1997 Nov;273(5):R1704-8. doi: 10.1152/ajpregu.1997.273.5.R1704. PMID 9374813
- [Background] Han DH, Hansen PA, Chen MM, Holloszy JO. DHEA treatment reduces fat accumulation and protects against insulin resistance in male rats. J Gerontol A Biol Sci Med Sci. 1998 Jan;53(1):B19-24. doi: 10.1093/gerona/53a.1.b19. PMID 9467418
- [Background] Villareal DT, Holloszy JO, Kohrt WM. Effects of DHEA replacement on bone mineral density and body composition in elderly women and men. Clin Endocrinol (Oxf). 2000 Nov;53(5):561-8. doi: 10.1046/j.1365-2265.2000.01131.x. PMID 11106916
- [Result] Villareal DT, Holloszy JO. Effect of DHEA on abdominal fat and insulin action in elderly women and men: a randomized controlled trial. JAMA. 2004 Nov 10;292(18):2243-8. doi: 10.1001/jama.292.18.2243. PMID 15536111